CLINICAL TRIAL: NCT01308372
Title: Cardiovascular Risk in General Practice in France
Brief Title: Cardiovascular Risk in General Practice in France: Cardiovascular Risk Week
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CFR-XXX-2011/1
Record Dates: First submitted 2011-02-18; First posted 2011-03-04 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: cardiovascular risk; France; General practice; Primary prevention; Non treated patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: For this group of patients, the cardiovascular risk will be evaluated by several tools: the SCORE scale, the Framingham 2008 scale d'Agostino and the 1998 scale Wilson ;

SUMMARY:
The purpose of this study is to evaluate the proportion of patients which present a high cardiovascular risk estimated by the SCORE scale, in general practice consultations of the 7 French regions (Paris area, North-East, Paris basin, West, South-West, South- East, Mediterranean area)

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* Without any personal history of coronary disease
* Non treated with lipid-lowering agents
* Lipid test = 1 year old
* Presenting at least one cardiovascular risk
* Visiting their General Practitioner

Exclusion Criteria:

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Probability Sample
Enrollment: 9246 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of cardiovascular risk in general practice in France estimated by the SCORE scale | 1 week

SECONDARY OUTCOMES:
Evaluation of cardiovascular risk in general practice in France estimated by the Framingham 2008 scale D'Agostino | 1 week
Evaluation of cardiovascular risk in general practice in France estimated by the Framingham 1998 scale Wilson | 1 week
Evaluation of arteries age evaluation by SCORE | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Eric BRUCKERT, Pr., Principal Investigator — Hôpital Pitié-Salpétrière - Service Endocrinologie-Métabolisme; Jean DALLONGEVILLE, Dr., Principal Investigator — Institut Pasteur de Lille - Unité d'Epidémiologie et de santé publique Inserm UMR 744; Jean FERRIERES, Pr., Principal Investigator — CHU Rangueil - Service de Cardiologie B - Toulouse; Serge KOWNATOR, Dr., Principal Investigator — Thionville -Société Française de Cardiologie
Locations (585):
- France (585):
  - Research Site, Achenheim, France
  - Research Site, Aizenay, France
  - Research Site, Albi, France
  - Research Site, Alençon, France
  - Research Site, Alès, France
  - Research Site, Algrange, France
  - Research Site, Alignan-du-Vent, France
  - Research Site, Allauch, France
  - Research Site, Alleins, France
  - Research Site, Allonnes, France
  - Research Site, Allouagne, France
  - Research Site, Ambès, France
  - Research Site, Ambleteuse, France
  - Research Site, Amelie Les Bains Palalda, France
  - Research Site, Amfreville, France
  - Research Site, Amiens, France
  - Research Site, Angers, France
  - Research Site, Aniche, France
  - Research Site, Annecy-le-Vieux, France
  - Research Site, Annemasse, France
  - Research Site, Annezin, France
  - Research Site, Annoeullin, France
  - Research Site, Anthony, France
  - Research Site, Antibes, France
  - Research Site, Anzin, France
  - Research Site, Arcachon, France
  - Research Site, Argeliers, France
  - Research Site, Argentan, France
  - Research Site, Armentières, France
  - Research Site, Arradon, France
  - Research Site, Arras, France
  - Research Site, Ars, France
  - Research Site, Asfeld, France
  - Research Site, Asnières-sur-Seine, France
  - Research Site, Aubagne, France
  - Research Site, Aubière, France
  - Research Site, Auchel, France
  - Research Site, Audincourt, France
  - Research Site, Auneau, France
  - Research Site, Aurillac, France
  - Research Site, Auxerre, France
  - Research Site, Avignon, France
  - Research Site, Avize, France
  - Research Site, Avord, France
  - Research Site, Avranches, France
  - Research Site, Badonviller, France
  - Research Site, Bailleul, France
  - Research Site, Bain-de-Bretagne, France
  - Research Site, Baixas, France
  - Research Site, Ballancourt, France
  - Research Site, Balma, France
  - Research Site, Bandol, France
  - Research Site, Banyuls de la Marenda, France
  - Research Site, Barbentane, France
  - Research Site, Basse-Goulaine, France
  - Research Site, Bassussarry, France
  - Research Site, Bazeilles, France
  - Research Site, Bazet, France
  - Research Site, Beaucouzé, France
  - Research Site, Beaumont-Hague, France
  - Research Site, Beaumont-lès-Valence, France
  - Research Site, Beaune-la-Rolande, France
  - Research Site, Beauvais, France
  - Research Site, Behren-lès-Forbach, France
  - Research Site, Belfort, France
  - Research Site, Belleville-sur-Meuse, France
  - Research Site, Bergerac, France
  - Research Site, Bernin, France
  - Research Site, Besançon, France
  - Research Site, Bessancourt, France
  - Research Site, Bétaille, France
  - Research Site, Bétheniville, France
  - Research Site, Béziers, France
  - Research Site, Biarritz, France
  - Research Site, Bitche, France
  - Research Site, Blagnac, France
  - Research Site, Blangy-sur-Bresle, France
  - Research Site, Blanzat, France
  - Research Site, Bléré, France
  - Research Site, Blois, France
  - Research Site, Boën-sur-Lignon, France
  - Research Site, Bois-Bernard, France
  - Research Site, Bolquère, France
  - Research Site, Bono, France
  - Research Site, Bonson, France
  - Research Site, Bordeaux, France
  - Research Site, Bosmie-l'Aiguille, France
  - Research Site, Bouguenais, France
  - Research Site, Bourbonne-les-Bains, France
  - Research Site, Bourg de Joué-sur-Erdre, France
  - Research Site, Bourges, France
  - Research Site, Bousse, France
  - Research Site, Boynes, France
  - Research Site, Brassac, France
  - Research Site, Bresles, France
  - Research Site, Brest, France
  - Research Site, Briançon, France
  - Research Site, Brie-Comte-Robert, France
  - Research Site, Bron, France
  - Research Site, Bruay-la-Buissière, France
  - Research Site, Bruay-sur-l'Escaut, France
  - Research Site, Cabannes, France
  - Research Site, Caen, France
  - Research Site, Cagnes-sur-Mer, France
  - Research Site, Cahagnes, France
  - Research Site, Calais, France
  - Research Site, Calonne-Ricouart, France
  - Research Site, Caluire-et-Cuire, France
  - Research Site, Cambrai, France
  - Research Site, Campagne-lès-Wardrecques, France
  - Research Site, Cancon, France
  - Research Site, Cannes, France
  - Research Site, Carnon-Plage, France
  - Research Site, Caromb, France
  - Research Site, Carpentras, France
  - Research Site, Carvin, France
  - Research Site, Castres, France
  - Research Site, Caudry, France
  - Research Site, Caunes-Minervois, France
  - Research Site, Cerizay, France
  - Research Site, Cessy, France
  - Research Site, Ceyrat, France
  - Research Site, Chambéry, France
  - Research Site, Champagne-sur-Oise, France
  - Research Site, Chanceaux-sur-Choisille, France
  - Research Site, Chaource, France
  - Research Site, Châlons-en-Champagne, France
  - Research Site, Châtillon-sur-Marne, France
  - Research Site, Chelles, France
  - Research Site, Chirac, France
  - Research Site, Claye-Souilly, France
  - Research Site, Clermont, France
  - Research Site, Clermont-Ferrand, France
  - Research Site, Clisson, France
  - Research Site, Clouange, France
  - Research Site, Collioure, France
  - Research Site, Colmar, France
  - Research Site, Colombey-les-Belles, France
  - Research Site, Colomiers, France
  - Research Site, Commercy, France
  - Research Site, Communay, France
  - Research Site, Cormeilles-en-Parisis, France
  - Research Site, Coudekerque-Branche, France
  - Research Site, Coulanges-la-Vineuse, France
  - Research Site, Courcelles-sur-Nied, France
  - Research Site, Cournon-d'Auvergne, France
  - Research Site, Coursan, France
  - Research Site, Crespin, France
  - Research Site, Crécy-en-Ponthieu, France
  - Research Site, Créhange, France
  - Research Site, Crêches-sur-Saône, France
  - Research Site, Cubjac, France
  - Research Site, Cucuron, France
  - Research Site, Cugnaux, France
  - Research Site, Dambach-la-Ville, France
  - Research Site, Danjoutin, France
  - Research Site, Denain, France
  - Research Site, Dessenheim, France
  - Research Site, Deuil-la-Barre, France
  - Research Site, Déville-lès-Rouen, France
  - Research Site, Diebling, France
  - Research Site, Dieppe, France
  - Research Site, Dijon, France
  - Research Site, Domène, France
  - Research Site, Domont, France
  - Research Site, Draguignan, France
  - Research Site, Dunières, France
  - Research Site, Einville-au-Jard, France
  - Research Site, Elliant, France
  - Research Site, Emmerin, France
  - Research Site, Eragny Sur Oise, France
  - Research Site, Excideuil, France
  - Research Site, Eyguières, France
  - Research Site, Échenoz-la-Méline, France
  - Research Site, Épinac, France
  - Research Site, Épinal, France
  - Research Site, Étampes-sur-Marne, France
  - Research Site, Évry, France
  - Research Site, Fegersheim, France
  - Research Site, Figeac, France
  - Research Site, Firminy, France
  - Research Site, Flavignac, France
  - Research Site, Fontaine-lès-Dijon, France
  - Research Site, Fontaine-Notre-Dame, France
  - Research Site, Fontenilles, France
  - Research Site, Fors, France
  - Research Site, Fos-sur-Mer, France
  - Research Site, Fosses, France
  - Research Site, Fraisses, France
  - Research Site, Francescas, France
  - Research Site, Frasne, France
  - Research Site, Fresnes-sur-Escaut, France
  - Research Site, Frontigny, France
  - Research Site, Frouard, France
  - Research Site, Gamaches, France
  - Research Site, Gap, France
  - Research Site, Gardanne, France
  - Research Site, Garges-lès-Gonesse, France
  - Research Site, Gerbéviller, France
  - Research Site, Gignac-la-Nerthe, France
  - Research Site, Givry-en-Argonne, France
  - Research Site, Gonesse, France
  - Research Site, Grasse, France
  - Research Site, Grenade-sur-l’Adour, France
  - Research Site, Grenoble, France
  - Research Site, Gréasque, France
  - Research Site, Grésy-sur-Aix, France
  - Research Site, Guesnain, France
  - Research Site, Guignicourt, France
  - Research Site, Guiscriff, France
  - Research Site, Guyancourt, France
  - Research Site, Hambye, France
  - Research Site, Hatten, France
  - Research Site, Hayange, France
  - Research Site, Hazebrouck, France
  - Research Site, Hellemmes-Lille, France
  - Research Site, Herblay-sur-Seine, France
  - Research Site, Herlies, France
  - Research Site, Héric, France
  - Research Site, Héricourt, France
  - Research Site, Holtzheim, France
  - Research Site, Hombourg, France
  - Research Site, Houilles, France
  - Research Site, Hyères, France
  - Research Site, Illkirch-Graffenstaden, France
  - Research Site, Issy-les-Moulineaux, France
  - Research Site, Ivry-sur-Seine, France
  - Research Site, Jardin, France
  - Research Site, Josnes, France
  - Research Site, Jouy-le-Châtel, France
  - Research Site, Juan-les-Pins, France
  - Research Site, Kurtzenhouse, France
  - Research Site, L'Haÿ-les-Roses, France
  - Research Site, L'Isle-sur-la-Sorgue, France
  - Research Site, La Boussac, France
  - Research Site, La Chabossière, France
  - Research Site, La Chaussée-Saint-Victor, France
  - Research Site, La Farlède, France
  - Research Site, La Forêt-sur-Sèvre, France
  - Research Site, La Garnache, France
  - Research Site, La Grand-Croix, France
  - Research Site, La Madeleine, France
  - Research Site, La Motte-Servolex, France
  - Research Site, La Neuville-Roy, France
  - Research Site, La Riche, France
  - Research Site, La Roche-en-Brenil, France
  - Research Site, La Rochelle, France
  - Research Site, La Saussaye, France
  - Research Site, La Teste-de-Buch, France
  - Research Site, La Tour-de-Salvagny, France
  - Research Site, La Turballe, France
  - Research Site, La Varenne-Saint-Hilaire, France
  - Research Site, Labouheyre, France
  - Research Site, Laguenne, France
  - Research Site, Lambersart, France
  - Research Site, Landeleau, France
  - Research Site, Landerneau, France
  - Research Site, Landrecies, France
  - Research Site, Langoiran, France
  - Research Site, Lapugnoy, France
  - Research Site, Lauzun, France
  - Research Site, Laval, France
  - Research Site, Lavardac, France
  - Research Site, Laventie, France
  - Research Site, Lavoûte-sur-Loire, France
  - Research Site, Laxou, France
  - Research Site, Lay-Saint-Christophe, France
  - Research Site, Le Bourget, France
  - Research Site, Le Cannet, France
  - Research Site, Le Clion-sur-Mer, France
  - Research Site, Le Gouray, France
  - Research Site, Le Grand-Lemps, France
  - Research Site, Le Grand-Quevilly, France
  - Research Site, Le Havre, France
  - Research Site, Le Houlme, France
  - Research Site, Le Lavandou, France
  - Research Site, Le Mée-sur-Seine, France
  - Research Site, Le Petit-Quevilly, France
  - Research Site, Le Pin-en-Mauges, France
  - Research Site, Le Plessis-Robinson, France
  - Research Site, Le Pontet, France
  - Research Site, Le Roc-Saint-André, France
  - Research Site, Le Russey, France
  - Research Site, Le Temple-de-Bretagne, France
  - Research Site, Le Vigan, France
  - Research Site, Lembach, France
  - Research Site, Les Clayes-sous-Bois, France
  - Research Site, Les Mureaux, France
  - Research Site, Les Pavillons-sous-Bois, France
  - Research Site, Les Sables-d'Olonne, France
  - Research Site, Levallois-Perret, France
  - Research Site, Liancourt, France
  - Research Site, Lieuran-lès-Béziers, France
  - Research Site, Liévin, France
  - Research Site, Lille, France
  - Research Site, Limoges, France
  - Research Site, Limoux, France
  - Research Site, Lingolsheim, France
  - Research Site, Lion-sur-Mer, France
  - Research Site, Loches, France
  - Research Site, Lodève, France
  - Research Site, Lomme, France
  - Research Site, Longpont-sur-Orge, France
  - Research Site, Longueau, France
  - Research Site, Loos-en-Gohelle, France
  - Research Site, Louviers, France
  - Research Site, Louvigny, France
  - Research Site, Lunéville, France
  - Research Site, Luxeuil-les-Bains, France
  - Research Site, Lœuilly, France
  - Research Site, Maché, France
  - Research Site, Magland, France
  - Research Site, Malakoff, France
  - Research Site, Malataverne, France
  - Research Site, Marcillé-Robert, France
  - Research Site, Margency, France
  - Research Site, Marignane, France
  - Research Site, Marles-les-Mines, France
  - Research Site, Maroilles, France
  - Research Site, Maromme, France
  - Research Site, Marquette-lez-Lille, France
  - Research Site, Marquion, France
  - Research Site, Marseille, France
  - Research Site, Marseillette, France
  - Research Site, Mauléon-Licharre, France
  - Research Site, Maxéville, France
  - Research Site, Meaux, France
  - Research Site, Mehun-sur-Yèvre, France
  - Research Site, Merlimont, France
  - Research Site, Merville, France
  - Research Site, Meslay-du-Maine, France
  - Research Site, Mesvres, France
  - Research Site, Metz, France
  - Research Site, Meylan, France
  - Research Site, Mélisey, France
  - Research Site, Méréville, France
  - Research Site, Mérignac, France
  - Research Site, Mézin, France
  - Research Site, Migniers, France
  - Research Site, Mions, France
  - Research Site, Molsheim, France
  - Research Site, Moncrabeau, France
  - Research Site, Monnières, France
  - Research Site, Montcenis, France
  - Research Site, Montdidier, France
  - Research Site, Montfaucon-Montigné, France
  - Research Site, Montfort-sur-Meu, France
  - Research Site, Montigny-le-Bretonneux, France
  - Research Site, Montluçon, France
  - Research Site, Montluel, France
  - Research Site, Montoir-de-Bretagne, France
  - Research Site, Montpellier, France
  - Research Site, Montreuil, France
  - Research Site, Montreuil-l'Argillé, France
  - Research Site, Montrond-le-Château, France
  - Research Site, Montrouge, France
  - Research Site, Morangis, France
  - Research Site, Moreuil, France
  - Research Site, Mougins Le Haut, France
  - Research Site, Mouilleron-le-Captif, France
  - Research Site, Mouliherne, France
  - Research Site, Moulins-lès-Metz, France
  - Research Site, Moutiers-les-Mauxfaits, France
  - Research Site, Mouvaux, France
  - Research Site, Mulhouse, France
  - Research Site, Mundolsheim, France
  - Research Site, Mûrs-Erigné, France
  - Research Site, Nalliers, France
  - Research Site, Nancy, France
  - Research Site, Nantes, France
  - Research Site, Narbonne, France
  - Research Site, Nasbinals, France
  - Research Site, Naucelle, France
  - Research Site, Neuilly-sur-Marne, France
  - Research Site, Neuilly-sur-Seine, France
  - Research Site, Nevers, France
  - Research Site, Nice, France
  - Research Site, Nieppe, France
  - Research Site, Nîmes, France
  - Research Site, Notre-Dame-d'Oé, France
  - Research Site, Notre-Dame-de-Monts, France
  - Research Site, Nouan-le-Fuzelier, France
  - Research Site, Noyon, France
  - Research Site, Oermingen, France
  - Research Site, Oignies, France
  - Research Site, Olivet, France
  - Research Site, Oradour-sur-Vayres, France
  - Research Site, Orchies, France
  - Research Site, Orléans, France
  - Research Site, Orthez, France
  - Research Site, Orvault, France
  - Research Site, Ostwald, France
  - Research Site, Paray-le-Monial, France
  - Research Site, Paris, France
  - Research Site, Parthenay, France
  - Research Site, Passy, France
  - Research Site, Pau, France
  - Research Site, Pauillac, France
  - Research Site, Pavilly, France
  - Research Site, Peltre, France
  - Research Site, Percy, France
  - Research Site, Pernes-les-Fontaines, France
  - Research Site, Perpignan, France
  - Research Site, Pessac, France
  - Research Site, Péronne, France
  - Research Site, Pfetterhouse, France
  - Research Site, Phalsbourg, France
  - Research Site, Pierrefitte-sur-Sauldre, France
  - Research Site, Pithiviers, France
  - Research Site, Pleubian, France
  - Research Site, Ploeren, France
  - Research Site, Plouzané, France
  - Research Site, Poissy, France
  - Research Site, Poitiers, France
  - Research Site, Pompey, France
  - Research Site, Pont-Aven, France
  - Research Site, Pont-à-Mousson, France
  - Research Site, Pont-de-l'Arche, France
  - Research Site, Portes-lès-Valence, France
  - Research Site, Pouilly-en-Auxois, France
  - Research Site, Pouilly-sous-Charlieu, France
  - Research Site, Puget-sur-Argens, France
  - Research Site, Puy-lÉvêque, France
  - Research Site, Puylaurens, France
  - Research Site, Puyricard, France
  - Research Site, Quarouble, France
  - Research Site, Quévreville-la-Poterie, France
  - Research Site, Quincy-Voisins, France
  - Research Site, Quint-Fonsegrives, France
  - Research Site, Ramonville-Saint-Agne, France
  - Research Site, Rauzan, France
  - Research Site, Râches, France
  - Research Site, Rebais, France
  - Research Site, Reims, France
  - Research Site, Renage, France
  - Research Site, Rennes, France
  - Research Site, Reyrieux, France
  - Research Site, Richebourg, France
  - Research Site, Richemont, France
  - Research Site, Riedisheim, France
  - Research Site, Rieux-Minervois, France
  - Research Site, Rigney, France
  - Research Site, Riom, France
  - Research Site, Rive-de-Gier, France
  - Research Site, Rognonas, France
  - Research Site, Romagnat, France
  - Research Site, Romagné, France
  - Research Site, Romainville, France
  - Research Site, Rosières-aux-Salines, France
  - Research Site, Roubaix, France
  - Research Site, Rouen, France
  - Research Site, Rousies, France
  - Research Site, Rouvroy, France
  - Research Site, Royan, France
  - Research Site, Rueil-Malmaison, France
  - Research Site, Rœulx, France
  - Research Site, Sail-sous-Couzan, France
  - Research Site, Sainghin-en-Mélantois, France
  - Research Site, Saint Maximin La Ste Baume, France
  - Research Site, Saint-Amant-Tallende, France
  - Research Site, Saint-Aubin-sur-Scie, France
  - Research Site, Saint-Barthélémy, France
  - Research Site, Saint-Bonnet-de-Mure, France
  - Research Site, Saint-Bonnet-le-Château, France
  - Research Site, Saint-Brieuc, France
  - Research Site, Saint-Chamond, France
  - Research Site, Saint-Claude-de-Diray, France
  - Research Site, Saint-Cyr-sur-Loire, France
  - Research Site, Saint-Denis-les-Ponts, France
  - Research Site, Saint-Denis-lès-Bourg, France
  - Research Site, Saint-Etienne, France
  - Research Site, Saint-Étienne-de-Montluc, France
  - Research Site, Saint-Étienne-du-Rouvray, France
  - Research Site, Saint-Étienne-lès-Remiremont, France
  - Research Site, Saint-Georges-de-Didonne, France
  - Research Site, Saint-Georges-du-Bois, France
  - Research Site, Saint-Germain-du-Puy, France
  - Research Site, Saint-Herblain, France
  - Research Site, Saint-Jean-de-Braye, France
  - Research Site, Saint-Jean-Pied-de-Port, France
  - Research Site, Saint-Julien-de-Civry, France
  - Research Site, Saint-Junien, France
  - Research Site, Saint-Laurent-de-Neste, France
  - Research Site, Saint-Laurent-du-Var, France
  - Research Site, Saint-Léger-des-Bois, France
  - Research Site, Saint-Léonard-de-Noblat, France
  - Research Site, Saint-Lô, France
  - Research Site, Saint-Martin-d'Oney, France
  - Research Site, Saint-Martin-la-Plaine, France
  - Research Site, Saint-Martin-le-Vinoux, France
  - Research Site, Saint-Maurice-lès-Châteauneuf, France
  - Research Site, Saint-Max, France
  - Research Site, Saint-Montan, France
  - Research Site, Saint-Nazaire, France
  - Research Site, Saint-Omer, France
  - Research Site, Saint-Orens-de-Gameville, France
  - Research Site, Saint-Ouen-du-Tilleul, France
  - Research Site, Saint-Pierre-des-Corps, France
  - Research Site, Saint-Priest, France
  - Research Site, Saint-Raphaël, France
  - Research Site, Saint-Saturnin-lès-Apt, France
  - Research Site, Saint-Sauflieu, France
  - Research Site, Saint-Savournin, France
  - Research Site, Saint-Victurnien, France
  - Research Site, Saint-Vincent-de-Tyrosse, France
  - Research Site, Saint-Vrain, France
  - Research Site, Samer, France
  - Research Site, Sarre-Union, France
  - Research Site, Sarrebourg, France
  - Research Site, Saverne, France
  - Research Site, Schiltigheim, France
  - Research Site, Schirrhein, France
  - Research Site, Segonzac, France
  - Research Site, Segré, France
  - Research Site, Senones, France
  - Research Site, Sessenheim, France
  - Research Site, Sevran, France
  - Research Site, Sète, France
  - Research Site, Sélestat, France
  - Research Site, Séné, France
  - Research Site, Six-Fours-les-Plages, France
  - Research Site, Sotteville-lès-Rouen, France
  - Research Site, Soucy, France
  - Research Site, St-Malo, France
  - Research Site, St.-Jean, France
  - Research Site, Stains, France
  - Research Site, Ste Anastasie, France
  - Research Site, Ste Feyre, France
  - Research Site, Ste Marguerite, France
  - Research Site, Ste Marie Aux Chenes, France
  - Research Site, Ste Savine, France
  - Research Site, Stiring-Wendel, France
  - Research Site, Strasbourg, France
  - Research Site, Sucé-sur-Erdre, France
  - Research Site, Surgères, France
  - Research Site, Tabanac, France
  - Research Site, Tarbes, France
  - Research Site, Targon, France
  - Research Site, Tarnos, France
  - Research Site, Taverny, France
  - Research Site, Terminiers, France
  - Research Site, Thiézac, France
  - Research Site, Toulouse, France
  - Research Site, Tourcoing, France
  - Research Site, Tours, France
  - Research Site, Tracy-le-Mont, France
  - Research Site, Troarn, France
  - Research Site, Valenciennes, France
  - Research Site, Vandœuvre-lès-Nancy, France
  - Research Site, Vannes, France
  - Research Site, Varennes-Vauzelles, France
  - Research Site, Vence, France
  - Research Site, Vendenheim, France
  - Research Site, Venelles, France
  - Research Site, Vernouillet, France
  - Research Site, Versailles, France
  - Research Site, Vertaizon, France
  - Research Site, Vélizy-Villacoublay, France
  - Research Site, Vémars, France
  - Research Site, Vic-la-Gardiole, France
  - Research Site, Vidauban, France
  - Research Site, Vieux-Condé, France
  - Research Site, Villefranche-sur-Saône, France
  - Research Site, Villefranque, France
  - Research Site, Villejuif, France
  - Research Site, Villeneuve-Loubet, France
  - Research Site, Villeneuve-sur-Lot, France
  - Research Site, Villeurbanne, France
  - Research Site, Villey-Saint-Étienne, France
  - Research Site, Villiers-en-Plaine, France
  - Research Site, Vitrolles, France
  - Research Site, Vitry-le-François, France
  - Research Site, Vittel, France
  - Research Site, Voiron, France
  - Research Site, Voisins-le-Bretonneux, France
  - Research Site, Voujeaucourt, France
  - Research Site, Wallers, France
  - Research Site, Warmeriville, France
  - Research Site, Wasquehal, France
  - Research Site, Wattrelos, France
  - Research Site, Waziers, France
  - Research Site, Willems, France
  - Research Site, Wingles, France
  - Research Site, Yenne, France
  - Research Site, Yutz, France